CLINICAL TRIAL: NCT00776555
Title: A Single-Blind, Randomized Study of the Comparative Drug Likeability and Pharmacokinetics of Vyvanse™ and ADDERALL XR® When Administered as a Solution
Brief Title: Compare Subjective Drug Liking & Pharmacokinetics of Vyvanse™ and ADDERALL XR® When Administered as an Oral Solution
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: The study was stopped by the sponsor based on a non-safety related business priority decision.
Sponsor: Shire (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: SPD489-112
Record Dates: First submitted 2008-10-20; First posted 2008-10-21 (Estimated); Results first posted 2010-07-07 (Estimated); Last update posted 2021-06-09 (Actual); Status verified 2021-05

CONDITIONS: Healthy
Keywords: Not required
MeSH Terms: interventions — Lisdexamfetamine Dimesylate

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Vyvanse™ (Experimental): 50mg capsule that has been emptied and made into solution
  Interventions: Drug: Lisdexamfetamine Dimesylate
- ADDERALL XR® (Experimental): 20mg capsule that has been emptied, crushed, and made into solution
  Interventions: Drug: Racemic mixture of dextroamphetamine and lisdexamfetamine

INTERVENTIONS:
Drug: Lisdexamfetamine Dimesylate — Study is a two-period cross-over design where subjects will have 2 Screening visits, a Baseline visit, and then be enrolled into the study for 2 Periods. Each Period has 2-3 visits and lasts from 2-6 weeks. At each Period visit subjects will be given one of the two treatment arm drugs that have been solubilized and then have blood drawn for pharmacokinetic analysis and the Drug Rating Questionnaire administered. At the end of Period 1 subjects will be crossed-over to the alternative treatment drug for the Period 2. The Vyvanse™ capsule contents will emptied into water to make a solution and given to subjects to drink at the beginning of each Period visit.
  Arms: Vyvanse™
Drug: Racemic mixture of dextroamphetamine and lisdexamfetamine — Same visits as described for Vyvanse™. The ADDERALL XR® capsule contents will be crushed, solubilized with water, and given to subjects to drink prior to pharmacokinetic blood draws and DRQ-S administration over the course of two periods.
  Arms: ADDERALL XR®

SUMMARY:
The purpose of this study is to compare subjective drug liking using the Drug Rating Questionnaire, subject version (DRQ-S), question 2 and pharmacokinetics of Vyvanse™ and ADDERALL XR® when administered as an oral solution.

Hypothesis: DRQ-S, question 2 will show no difference between the two drugs

DETAILED DESCRIPTION:
Not required

ELIGIBILITY:
Inclusion Criteria

* Healthy young adults, male or female (non-pregnant and non-lactating), age 18-25 years at time of consent
* Have a body mass index (BMI) between 20.0 and 29.0kg/m2
* Satisfactory medical assessment with no clinically significant or relevant
* Subject must demonstrate a positive response to amphetamine at Screening

Exclusion Criteria

* A history of current or recurrent disease that could have an effect on the study
* Subject has a history of seizures, any tic disorder, or a current diagnosis and/or a known family history of Tourette's Disorder
* Subject has a concurrent chronic or acute illness or other condition that might confound the results of safety assessments or that might increase risk to the subject
* Subject has any clinically significant ECG and/or laboratory abnormalities
* Subject has a documented allergy, hypersensitivity or intolerance to amphetamines
* Subject has been prescribed or has taken amphetamine products in the past, including childhood; recreational use may not be exclusionary per the Investigator's discretion
* Subject has a known family history of sudden cardiac death or ventricular arrhythmia
* Subject has a recent history (within the past 6 months) of suspected substance abuse or dependence disorder (excluding nicotine)
* Subject has participated in any investigational clinical or vaccine trial within 30 days prior to the first dose of study drug
* Subjects is currently considered a suicide risk, has previously made a suicide attempt or has a prior history of, or is currently demonstrating suicidal ideation

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 3 (Actual)
Dates: Start 2008-11-21 (Actual); Primary Completion 2009-03-31 (Actual); Study Completion 2009-03-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Shire decided to cancel this study on march 31, 2009 due to changes in business priorities. The study termination was not related to any data or safety concerns.
Groups:
- Vyvanse First: Vyvanse 50mg capsule that has been emptied and made into an oral solution in first intervention, washout, then Adderall XR20mg capsule that has been emptied, crushed, and made into an oral solution in second intervention
- ADDERALL XR First: Adderall XR 20mg capsule that has been emptied, crushed, and made into an oral solution in the first intervention, washout, then Vyvanse 50mg capsule that has been emptied and made into an oral solution in second intervention
Period: Overall Study
Arm/Group | Vyvanse First | ADDERALL XR First
Started | 3 | 0
Completed | 0 | 0
Not Completed | 3 | 0
Not completed — Study terminated | 3 | 0

BASELINE CHARACTERISTICS:
Population: At the time of the premature study termination, only 3 participants had been enrolled into this study. All 3 participants were randomized to receive VYVANSE in Period 1 of this study, and ADDERALL XR in Period 2 of this study. None of the study participants advanced to Period 2, therefore none received ADDERALL XR.
Groups:
- Total: Total of all reporting groups
Arm/Group | Vyvanse First | ADDERALL XR First | Total
Number analyzed (Participants) | 3 | 0 | 3
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 |  | 0
  Between 18 and 65 years | 3 |  | 3
  >=65 years | 0 |  | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 |  | 1
  Male | 2 |  | 2
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 3 |  | 3

OUTCOME MEASURES:

1. Primary Outcome: Drug Rating Questionnaire-Subject (DRQ-S), Question 2
Description: Question 2: How much do you like the effects you are feeling now? Questions are rated on a 29-point scale from 1 (not at all) to 29 (an awful lot). The higher the score the stronger the subjective experience. This is a subjective measure of a drug's effect that has been used to assess the abuse potential of drugs.
Time Frame: Pre-dose and 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 7, 8, 12 and 24 hours post-dose
Population: Analysis not performed because of the study's premature termination.
Arm/Group | Vyvanse First | ADDERALL XR First
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: DRQ-S, Question 1
Description: Question 1: How much do you feel the drug now? Questions are rated on a 29-point scale from 1 (not at all) to 29 (an awful lot). The higher the score the stronger the subjective experience. This is a subjective measure of a drug's effect that has been used to assess the abuse potential of drugs.
Time Frame: Pre-dose and 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 7, 8, 12 and 24 hours post-dose
Population: Analysis not performed because of the study's premature termination.
Arm/Group | Vyvanse First | ADDERALL XR First
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: DRQ-S, Question 3
Description: Question 3: Do you dislike the drug effect you are feeling now? Questions are rated on a 29-point scale from 1 (not at all) to 29 (an awful lot). The higher the score the stronger the subjective experience. This is a subjective measure of a drug's effect that has been used to assess the abuse potential of drugs.
Time Frame: Pre-dose and 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 7, 8, 12 and 24 hours post-dose
Population: Analysis not performed because of the study's premature termination.
Arm/Group | Vyvanse First | ADDERALL XR First
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Shire decided to cancel this study on march 31, 2009 due to changes in business priorities. The study termination was not related to any data or safety concerns.
Description: Note: At the time of the premature termination, only 3 participants had been enrolled into this study. All 3 participants were randomized to receive VYVANSE in Period 1 of this study, and ADDERALL XR in Period 2 of this study. None of the study participants advanced to Period 2, therefore none received ADDERALL XR.
Arm/Group | Vyvanse First | ADDERALL XR First
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/0
Other Adverse Events (participants affected / at risk) | 2/3 | 0/0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Vyvanse First (N=3) | ADDERALL XR First (N=0)
Headache (Nervous system disorders) | 1 | 0
Upper respiratory infection (Infections and infestations) | 1 | 0

LIMITATIONS AND CAVEATS:
Shire decided to cancel this study on march 31, 2009 due to changes in business priorities. The study termination was not related to any data or safety concerns.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If a multicenter publication is not submitted within twelve (12) months after conclusion, abandonment or termination of the Study at all sites, or after Sponsor confirms there shall be no multicenter Study publication, the Institution and/or such Principal Investigator may publish the results from the Institution site individually.